CLINICAL TRIAL: NCT00038519
Title: An Open Label, Phase II Study of Amprenavir/Ritonavir or Saquinavir/Ritonavir in HIV-Infected Subjects Following Failure With Kaletra (Lopinavir/Ritonavir) as Their Second Protease Inhibitor.
Brief Title: Amprenavir/Ritonavir or Saquinavir/Ritonavir in HIV-Infected Subjects Following Failure With Kaletra as Their Second Protease Inhibitor
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M00-261
Record Dates: First submitted 2002-05-31; First posted 2002-06-03 (Estimated); Last update posted 2006-07-28 (Estimated); Status verified 2006-07

CONDITIONS: HIV Infections
Keywords: treatment experienced; HIV
MeSH Terms: conditions — HIV Infections | interventions — amprenavir; Ritonavir; Saquinavir

INTERVENTIONS:
Drug: Amprenavir/ritonavir
Drug: Saquinavir/ritonavir

SUMMARY:
The purpose of this study is to study the safety and efficacy of Amprenavir/ritonavir or saquinavir/ritonavir in HIV infected patients that have failed Kaletra as their second protease inhibitor based HAART.

ELIGIBILITY:
Inclusion:

* Subject must remain on current antiretroviral therapy during screening until a new regimen is initiated.
* Subject demonstrates reduced susceptibility to lopinavir.
* Subject's two most recent viral loads obtained after at least 16 weeks of lopinavir/ritonavir therapy, and while still on Kaletra therapy must be at least 1,000 copies/mL.
* The Kaletra regimen must be the subject's second PI containing regimen and must not contain any other PIs.
* Subject is at least 18 years of age.
* Subject has not been treated for an active opportunistic infection within 30 days of screening.

Exclusion:

* Subject has a history of active substance abuse or psychiatric illness that could preclude compliance to the protocol.
* Female subject pregnant or lactating.
* Use of an Investigational drug within 30 days prior to the initiation of drug dosing.
* Subject is receiving systemic chemotherapy.
* Subject has a history of acute or chronic pancreatitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16
Dates: Start 2001-04

PRIMARY OUTCOMES:
Proportion of subjects with plasma HIV RNA levels below the limit of quantification (400 copies/mL) at week 24 and the time until loss of virologic response through week 48

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Sun, M.D., Study Chair — Divisional Vice President, Infectious Diseases and Virology Development
Locations (52):
- United States (23):
  - Phoenix Body Positive, Inc., Phoenix, Arizona
  - AIDS Health Care Foundation - Research Center, Los Angeles, California
  - 20th Avenue Medical Center Kaiser Permanente, Denver, Colorado
  - University of Colorado Health Sciences Center, Denver, Colorado
  - IDC Research Initiative, Altamonte Springs, Florida
  - Gary J. Richmond, M.D., Fort Lauderdale, Florida
  - Associates in Research, Fort Myers, Florida
  - University of Miami School of Medicine, Miami, Florida
  - Infectious Disease Research Institute, Inc., Tampa, Florida
  - AIDS Research Consortium of Atlanta, Inc., Atlanta, Georgia
  - CORE Center, Chicago, Illinois
  - Donna E. Sweet, M.D., Wichita, Kansas
  - David Parks, M.D., St Louis, Missouri
  - Saint Michael's Medical Center, Newark, New Jersey
  - Howard A. Grossman, M.D., New York, New York
  - John B. Montana, M.D., New York, New York
  - State University of New York at Stony Brook, Stony Brook, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - The Research & Education Group, Portland, Oregon
  - Bornemann Internal Medicine, Reading, Pennsylvania
  - David Wright, M.D., Austin, Texas
  - Diversified Medical Practices, P.A., Houston, Texas
  - Hampton Roads Medical Specialists, Hampton, Virginia
- Argentina (2):
  - Hospital Muniz - FUNDAI, Buenos Aires
  - Fundacion Huesped, Buenos Aires
- Brazil (3):
  - Hospital do Servidor Publico Estadual de Sao Paulo, São Paulo, São Paulo
  - Hospital Evandro Chagas - Fiocryz, Rio de Janeiro
  - Hospital Heliopolis, São Paulo
- Canada (4):
  - Phillip Sestak, M.D, Vancouver, British Columbia
  - Ottawa Hospital General Campus, Ottawa, Ontario
  - Toronto General Hospital Division of The University Health Network, Toronto, Ontario
  - Montreal Chest Institute/Royal Victoria Hospital, Montreal, Quebec
- France (6):
  - Tour Drouet - C.H.U. Brabois, Vandœuvre-lès-Nancy, Cedex
  - Service du C.I.S.I.H. - C.H.U. de Grenoble, La Tronche
  - Hospital Tenon, Paris
  - Groupe Hospitalier Cochin -Saint-Vincent-de-Paul La Roche-Guyon, Paris
  - Hospital Yves Le Foll, Saint-Brieuc
  - La Seyne sur Mer, Hopital Chalucet, Toulon
- Italy (4):
  - S. Raffaele Hospital, Milan
  - III Infectious Diseases Division IRCCS "L. Spallanzani", Rome
  - IRCCS "L. Spallanzani", Rome
  - Hospital "Amedeo di Savoia", Torino
- Wojewodzki Szpital Zakazny, Warsaw, Poland
- Puerto Rico (2):
  - Centro Familiar, Inc, Ponce
  - New Puerto Rico CONCRA, Rio Piedras
- Spain (6):
  - Hospital Germans Trias I Pujol, Badalona
  - Hospital De La Sta Creu I San Pau, Barcelona
  - Hospital Clinic I Provincial, Barcelona
  - Hospital Carlos III, Madrid
  - Hospital La Paz, Madrid
  - Hospital Universitario Vergen del Rocio, Seville
- Royal Free Hospital, London, United Kingdom